CLINICAL TRIAL: NCT00270816
Title: Effect of Cyclical Administration of Interferon β-1b in Multiple Sclerosis - Comparison With Normal Dose.
Brief Title: Interferon ß-1b Treatment by Cyclical Administration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: S. Andrea Hospital (Other)
Collaborators: Italian Multiple Sclerosis Foundation (Other)
Responsible Party: Principal Investigator, Giovanni Ristori, MD, S. Andrea Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU - CYC - 06
Record Dates: First submitted 2005-12-27; First posted 2005-12-28 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Interferon-ß-1b; Therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interferon beta cyclical administration (Experimental): Interferon ß-1b Treatment by Cyclical Administration
  Interventions: Drug: Interferon-ß-1b
- Interferon ß-1b Treatment (Active Comparator): Interferon ß-1b Treatment
  Interventions: Drug: Interferon ß-1b

INTERVENTIONS:
Drug: Interferon-ß-1b — 250 micrograms (8 MIU) administered subcutaneously (sc) every other day with a discontinuance month every 2 months
  Arms: interferon beta cyclical administration
Drug: Interferon ß-1b — 250 micrograms (8 MIU) administered subcutaneously (sc) every other day
  Arms: Interferon ß-1b Treatment

SUMMARY:
The therapy with Interferon-ß-1b reduces the inflammatory component of multiple sclerosis with positive effects on the disease course. The 8 MUI dose at alternate days is kept constant for years. About 1/3 of patients suspend treatment by three years due to side effects or suspected or accepted ineffectiveness. The main objective of the study is to verify the safety and effectiveness of a cyclical administration (a month of suspension after two of treatment) from the beginning of treatment. There is the possibility that a scheme envisaging therapy free intervals can reduce the onset of negative feedbacks (antagonising the drug therapeutic effect) compared to the standard administration protocol. This might also result in an increase of the drug effectiveness and/or in a longer duration of effectiveness itself. Finally, cyclical administration allows patients to spend actual periods of "therapeutic vacation", with positive psychological effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by remitting Multiple Sclerosis who had at least a relapse in the last year of the disease.
* Satisfying general clinical conditions according to the researcher. Adequate hepatic function. Capacity to use adequate contraceptive techniques during the study.

Exclusion Criteria:

* Any other disease that might better explain signs and symptoms of the patient.
* Any other disability condition that might interfere with the clinical evolution.
* History of hypersensitivity to natural or recombinant interferon or to human albumin.
* Clinically significant heart diseases and not controlled like dysrhythmias, angina pectoris or congestive heart failure.
* Not adequately controlled epilepsy.
* Inability, according to the examining commission, to grant a complete compliance with the protocol requirements for the whole study.
* Previous therapies modifying the disease course in the last six months.
* Steroid therapies in the last 3 months.
* Pregnancy, lactation, serological positivity to the pregnancy test during the screening period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
number of gad-enhancing lesions (CELs) in T1 | baseline and after 12 months
  Group (cyclic withdrawal vs full regimen) differences in the cumulative number of CELs

SECONDARY OUTCOMES:
number of new and enlarging T2 lesions | baseline and after 12 months
  Group (cyclic withdrawal vs full regimen) differences in new and enlarging T2 lesions
volume of T1 lesions (black holes) | baseline and after 12 months
  Group (cyclic withdrawal vs full regimen) differences in T1 lesion volume (black holes)
relapse rate | baseline and after 12 months
  Group (cyclic withdrawal vs full regimen) differences in relapse rate

CONTACTS AND LOCATIONS:
Overall Officials: Marco Salvetti, MD, Study Director — S.Andrea Hospital, University of Rome "La Sapienza"
Locations (1):
- Azienda Ospedaliera S. Andrea, II Facoltà di Medicina e Chirurgia, Università di Roma "La Sapienza", Rome, Italy

REFERENCES:
- [Background] Steinman L. Immunotherapy of multiple sclerosis: the end of the beginning. Curr Opin Immunol. 2001 Oct;13(5):597-600. doi: 10.1016/s0952-7915(00)00266-1. PMID 11544011
- [Background] Calabresi PA, Stone LA, Bash CN, Frank JA, McFarland HF. Interferon beta results in immediate reduction of contrast-enhanced MRI lesions in multiple sclerosis patients followed by weekly MRI. Neurology. 1997 May;48(5):1446-8. doi: 10.1212/wnl.48.5.1446. PMID 9153489
- [Background] Richert ND, Zierak MC, Bash CN, Lewis BK, McFarland HF, Frank JA. MRI and clinical activity in MS patients after terminating treatment with interferon beta-1b. Mult Scler. 2000 Apr;6(2):86-90. doi: 10.1177/135245850000600206. PMID 10773853
- [Background] Langenkamp A, Messi M, Lanzavecchia A, Sallusto F. Kinetics of dendritic cell activation: impact on priming of TH1, TH2 and nonpolarized T cells. Nat Immunol. 2000 Oct;1(4):311-6. doi: 10.1038/79758. PMID 11017102
- [Background] Rissoan MC, Soumelis V, Kadowaki N, Grouard G, Briere F, de Waal Malefyt R, Liu YJ. Reciprocal control of T helper cell and dendritic cell differentiation. Science. 1999 Feb 19;283(5405):1183-6. doi: 10.1126/science.283.5405.1183. PMID 10024247
- [Background] Skok J, Poudrier J, Gray D. Dendritic cell-derived IL-12 promotes B cell induction of Th2 differentiation: a feedback regulation of Th1 development. J Immunol. 1999 Oct 15;163(8):4284-91. PMID 10510367
- [Background] McDonald WI, Compston A, Edan G, Goodkin D, Hartung HP, Lublin FD, McFarland HF, Paty DW, Polman CH, Reingold SC, Sandberg-Wollheim M, Sibley W, Thompson A, van den Noort S, Weinshenker BY, Wolinsky JS. Recommended diagnostic criteria for multiple sclerosis: guidelines from the International Panel on the diagnosis of multiple sclerosis. Ann Neurol. 2001 Jul;50(1):121-7. doi: 10.1002/ana.1032. PMID 11456302
- [Background] Pozzilli C, Bastianello S, Koudriavtseva T, Gasperini C, Bozzao A, Millefiorini E, Galgani S, Buttinelli C, Perciaccante G, Piazza G, Bozzao L, Fieschi C. Magnetic resonance imaging changes with recombinant human interferon-beta-1a: a short term study in relapsing-remitting multiple sclerosis. J Neurol Neurosurg Psychiatry. 1996 Sep;61(3):251-8. doi: 10.1136/jnnp.61.3.251. PMID 8795595
- [Derived] Romano S, Ferraldeschi M, Bagnato F, Mechelli R, Morena E, Caldano M, Buscarinu MC, Fornasiero A, Frontoni M, Nociti V, Mirabella M, Mayer F, Bertolotto A, Pozzilli C, Vanacore N, Salvetti M, Ristori G. Drug Holiday of Interferon Beta 1b in Multiple Sclerosis: A Pilot, Randomized, Single Blind Study of Non-inferiority. Front Neurol. 2019 Jul 16;10:695. doi: 10.3389/fneur.2019.00695. eCollection 2019. PMID 31379701
- See also: SPONSOR SITE — http://www.ospedalesantandrea.it